CLINICAL TRIAL: NCT02609516
Title: What is the Impact of Socioeconomic Inequalities in the Rates of Transition Between Health, Multimorbidity and Death Amongst Older People in England?
Brief Title: Impact of Socioeconomic Inequalities in Transition Between Health, Multimorbidity and Death Amongst Older People
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Harry Hemingway, Professor of Epidemiology and Public Health, University College, London
Other Study IDs: 14_179
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Multimorbidity
Keywords: Multimorbidity; Health inequalities; Ageing; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy: Patients without any of the pre-specified chronic diseases
  Interventions: Other: This is not an intervention study
- Multimorbid: Patients having any two or more of the pre-specified chronic diseases
  Interventions: Other: This is not an intervention study

INTERVENTIONS:
Other: This is not an intervention study — This study is based on the retrospective analysis of linked electronic health records.

SUMMARY:
Life expectancy at age 65 in the most deprived fifth of the English population was about 4 years shorter than of the most affluent fifth in 2010. The inverse gradient between mortality and social position is well established. But how disease patterns and multimorbidity (having two or more long term conditions at the same time) impact on differential mortality rates is inconclusive: is it because disadvantaged groups acquire more or more lethal combinations of, diseases over their life course; or, simply, become ill at ages younger than more affluent groups?

DETAILED DESCRIPTION:
The association between social inequality and cause-specific mortality and single disease morbidity has been studied extensively. However, it remains unclear whether having two or more chronic diseases concurrently (or 'multimorbidity') plays a role in contributing to the inequalities gap in survival. This is particularly relevant given an ageing population and the trend of a widening in the life expectancy gap across several European countries.

Multimorbidity incidence increases rapidly with age. Estimates of the prevalence of multimorbidity in older people range from 55% to 98%, mainly due to the selection of diseases included, population coverage (hospital, community) and data source (self-reported surveys or clinical records). However, across all studies there is a clear and consistent pattern of higher prevalence rates at older ages, with multimorbidity.

Many aspects of the patient health trajectory remain under-explored. Patient case-mixes are likely to vary across socioeconomic groups, alongside a host of prognostic factors, including the clustering of multiple risk factors, age of onset, and disease presentation, progression and management in the presence of multiple health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Registered with a participating practice that has agreed to data linkage
* Registered with an 'up to standard' participating general practice for at least 1 year
* Aged 45 and over on Jan 1st 2001 or who turn 45 between 1st Jan 2001 and 25th March 2010, irrespective of initial health status.

Exclusion Criteria:

* Patients with a record unlinked to deprivation due to missing or incomplete postcode of residence.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients included in the CALIBER dataset.
Sampling Method: Non-Probability Sample
Enrollment: 1300000 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Yearly multimorbidity incidence rate | 10 years
  Numerator: Of patients with either 0 or 1 chronic diseases as on 1st Jan of the year, all those who become multimorbid by 31st Dec of the year.
  Denominator: patient years at risk of patients with either 0 or 1 chronic diseases as on 1st Jan of the year
Yearly multimorbidity prevalence | 10 years
  Numerator: all those with 2 or more listed diseases on 1st July of the year. Denominator: All eligible patients on 1st July of the year, irrespective of disease status on that date.
Yearly all-cause mortality rates | 10 years
  Numerator: number of deaths until 31st Dec of the year amongst the patients included in the denominator.
  Denominator: Person years at risk of patients with 0,1,2 or more diseases on 1st Jan of the year.
Overall life expectancy | 10 years
  Incident rates of transitions between no disease, 1 disease, 2+ diseases, and death.
Health state-specific life expectancies | 10 years
  Incident rates of transitions between four health states - no disease, 1 disease, 2+ diseases, and death.

SECONDARY OUTCOMES:
Yearly non-accidental mortality rates | 10 years
  As outcome 3 but excluding accidental deaths from the numerator

CONTACTS AND LOCATIONS:
Overall Officials: Madhavi Bajekal, PhD, Study Director — University College, London
Locations (1):
- University College London, London, United Kingdom